CLINICAL TRIAL: NCT04795401
Title: The Effectiveness of FRAME FR for ArterioVenous Fistula Repair in High-Flow Reduction, A Prospective, Monocenter Controlled Trial
Brief Title: The Effectiveness of FRAME FR for AVF Repair in High-Flow Reduction & Stabilization, A Prospective Trial
Acronym: FRAME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRAME-FR
Record Dates: First submitted 2021-02-22; First posted 2021-03-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Arteriovenous Fistula
Keywords: Arteriovenous Fistula; Fistula reconstruction
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FRAME Group (Experimental): Patients will be enrolled during their hospitalization/consultation in vascular surgery department. After asking questions, his given free, informed and written consent will be collected, and recorded in his medical file by the investigator.
  During this hospitalization, the pre-procedure forming part of the usual care is carried out. The specific acts of research are: Cardiac echocardiography and Quality of life survey SF-36 The plication procedure will be performed according to the FRAME FR. All pre-, peri-, and post- operative routine patient management will be carried out as usual.
  Follow up visits will be held at 6, 12 months post procedure. All follow up visits will include the assessments as usual.
  The specific acts of research are as follows: Cardiac echocardiography at 12 months and quality of life survey SF-36.
  Interventions: Device: FRAME FR IFU
- Control Group (No Intervention): Control group corresponds to the historical patients over a period of time sufficient to have at least 20 patients according to inclusion criteria. The information form will be sent to each patient eligible for the study by post. Without any feedback from him within 30 days, it is considered that the patient does not object to the use of its data.
  As part of this research, no additional examination will be performed. The data used correspond to the data collected in the usual care of patients.

INTERVENTIONS:
Device: FRAME FR IFU — The surgeon will use the medical device FRAME to perform the plication procedure. The device will be selected and implanted according to the product IFU.
  Arms: FRAME Group

SUMMARY:
Patients with end-stage renal disease require permanent vascular access to enable safe and effective hemodialysis. An arteriovenous fistula (AVF), where a vein is mobilized and connected to an artery in the arm, is considered the gold standard and first choice for vascular access. After fistula creation, the vein is subjected to high pressure and flow, and undergoes remodeling. This includes the possibility of significant dilatation and intimal hyperplasia. Normal AVF flow required for effective dialysis is around 0.6 liters/min or 0.4-0.8 liters/min. However, in at least 20% of patients, excessive remodeling and dilatation of the fistula result in a high flow AVF with >2 liters/min.

High flow fistulas significantly increase the risk for the development of high output cardiac failure, skin breakdown, bleeding, hand ischemia, and other systemic complications. In cases of high flow AVF, venous reconstruction procedures, banding and/or plication, are often required to limit venous diameter and flow. The longevity of this procedure is limited as the reconstructed segment remodels and re-dilates due to ongoing arterial pressure. Banding and plication are both procedures that are designed to increase resistance to flow. Banding is performed by wrapping a segment of polytetrafluoroethylene (PTFE) around the outflow tract of the fistula, or by placing a suture around the fistula near the arterial anastomotic area to create a narrowing. Fistula plication involves narrowing of a short segment of the proximal venous outflow tract, usually accomplished by suturing or stapling the fistula for 2-6 cm. One of the notable systemic effects of a hemodialysis AVF is an acute decrease in systemic vascular resistance with a simultaneous increase in venous return to the heart, and thus an increase of the cardiac output. Cardiac failure occurs more frequently in patients with an access flow QA>2 l/min and CPR≥20%. Another adverse systemic effect of AV fistulas is pulmonary hypertension. The increased flow volume to the heart from an AV fistula yields an increase in pulmonary pressures. This can limit pulmonary vasodilation and result in pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* Patient with a fistula flow >1.5l/min
* Patient with a hemodialysis AVF and heart failure symptoms and who may require a reduction in flow even if <1.5l/min
* Patient whose AVF flows <1.5l/min and who may require a flow reduction for a reduction of edema in case of central vein stenosis or symptom of steal syndrome
* Patient referred by a cardiologist for high output cardiac failure
* Patient who is able and willing to comply with the study follow up requirements
* French speaking patient
* Patient who is affiliated to a social security system
* Patient who is able and willing to give his informed written consent.

Exclusion Criteria:

* Patient with any local near fistula or systemic sign or infection
* Patient with AV Fistula composite (constructed or prosthetic graft and vein
* Patient with stents within the operative portion of the fistula
* Patients with known central venous stenosis or occlusion
* Patients with a hand ischemia
* Patient with wall thickness >2 mm, with separation or thrombus within the operative portion of the fistula that cannot be removed, as determined intraoperatively
* Hypercoagulability, on chronic anticoagulation
* Pregnant and breastfeeding women
* Concomitant life-threatening disease, likely to limit life expectancy to less than two years
* Inability to tolerate or comply with required guideline based upon post-operative drug regimen
* Inability to tolerate or comply with required follow-ups
* Concurrent participation in an interventional (drug or device) study for which the follow-up is not completed
* Patient unable or unwilling to perform all the requested tasks
* Patient under tutorship or curatorship
* Patient deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Fistula flow Evaluation M6 | Month 6
  The primary outcome of the research is to evaluate the fistula flow by Doppler Us and the fistula primary patency rate over time.
Fistula flow Evaluation M12 | Month12
  The primary outcome of the research is to evaluate the fistula flow by Doppler Us and the fistula primary patency rate over time

SECONDARY OUTCOMES:
Occurence of safety events | at 6 and 12 months
  This outcome corresponds to the number of safety events such as death, infection, ongoing steal, recurrent aneurysm, new cephalic arch stenosis, fistula thrombosis.
Evaluation of the functional fistula patency | at 6 and 12 months
  This ouctome corresponds to functional fistula patency.
Cardiac parameters | at 12 months
  CPR = QA/CO ratio
Secondary patency | at 6 and 12 months
  This outcome corresponds to the evaluation of thrombosis and AVF discontinuation at 6 and 12 months.
Patient's Quality of Life SF-36 | at 6 and 12 months
  The SF-36 questionnaire consists of 36 items, which are used to calculate eight subscales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). The first four scores can be summed to create the physical composite score (PCS), while the last four can be summed to create the mental composite score (MCS). Scores for the SF-36 scales range between 0 and 100, with higher scores indicating a better HRQOL.
Reintervention | at 6 and 12 months
  This outcome is to evaluate the number of patients who had a surgical or endovascular reintervention at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros MALLIOS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- See also: Amerling et al. Arteriovenous Fistula Toxicity. Blood Purif 2011; 31: 113-120. — https://pubmed.ncbi.nlm.nih.gov/21228578/
- See also: Sheaffer et al. Minimally Invasive Limited Ligation Endoluminal-Assisted Revision (MILLER): A Review of the Available Literature and Brief Overview of Alternate Therapies in Dialysis Associated Steal Syndrome. J. Clin. Med. 2018, 7, 128. — https://pubmed.ncbi.nlm.nih.gov/29843483/
- See also: Reddy YNV, Obokata M, Dean PG, et al. Long-term cardiovascular changes following creation of arteriovenous fistula in patients with end stage renal disease. Eur Heart J 2017; 38:1913 — https://pubmed.ncbi.nlm.nih.gov/28329100/
- See also: Basile et al. The relationship between the flow of arteriovenous fistula and cardiac output in haemodialysis patients — https://pubmed.ncbi.nlm.nih.gov/17942475/